CLINICAL TRIAL: NCT06081439
Title: Validating Immunological Markers in Blood and Cerebrospinal Fluid Associated With Mental Fatigue in Graves' Disease and Their Association With Functional Changes in Neuronal Activation
Brief Title: Validating Immunological Markers Associated With Mental Fatigue in Graves' Disease
Status: Recruiting | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: ImmunoGraves wp2
Record Dates: First submitted 2023-09-28; First posted 2023-10-13 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Graves Disease; Mental Fatigue
MeSH Terms: conditions — Graves Disease; Mental Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients: 310
- controls: 120

SUMMARY:
Mental fatigue occurs in many diseases and the reasons are mostly unknown. The investigators hypothesize that remaining mental fatigue after restored euthyroidism in Graves' disease is an autoimmune complication. This is a confirmatory study of the biomarkers from ImmunoGraves WP1 in which immunological markers with possible association with mental fatigue in Graves' disease are explored.

In ImmunoGraves WP2, 310 patients with Graves' disease are assessed for symptoms of mental fatigue, quality of life, anxiety and depression, self-evaluated stress, coping strategies, personality traits, eye symptoms and background variables. Participants are examined in hyperthyroidism at inclusion, within three weeks from diagnosis, and in euthyroidism after 15 months. Serum and cerebrospinal fluid (in a subsample of participants) is collected at both visits and will be evaluated for the immunological markers identified in WP1 as well as for thyroid hormones, thyroid autoantibodies and biomarkers indicating organic and structural nerve damage. Significant predictors for mental fatigue will be identified by logistic regression.

To assess functional changes in the brain, magnetoencephalography will be performed in a subset of patients and in healthy controls at inclusion and after 15 to 18 months. Combined with magneto resonance imaging (MRI), magnetoencephalography gives information on neuronal activation during attention testing.

ELIGIBILITY:
Inclusion Criteria:

* Recently diagnosed Graves' disease
* Positive thyroid stimulating hormone (TSH)-receptor antibodies (TRAb)
* Thyroid hormones above the upper reference limit
* Inclusion within three weeks after start of antithyroid drugs

Controls: Matched for gender and age

Exclusion Criteria:

* Person unable to follow protocol as with psychosis, dementia or not able to answer questionnaires in Swedish.
* Recidive of Graves' disease
* Pregnancy

Controls: -Thyroid disease

* Neurological disease

Ages: 18 Years to 72 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 310 patients with Graves' are recruited from Endocrine Clinic at Sahlgrenska University Hospital and Östra Hospital. Patients meeting the inclusion criteria are consecutively asked to participate. A subgroup of maximum 120 patients who are willing to give cerebrospinal fluid are recruited to the sub-study with magnetoencephalography. Controls to this sub-study are recruited from records from the tax authority.
Sampling Method: Probability Sample
Enrollment: 430 (Estimated)
Dates: Start 2019-09-12 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Identifying the immunological markers in blood at inclusion that significantly increases the risk for mental fatigue at follow up. | Blood drawn at inclusion. Mental Fatigue Scale completed by participants at follow-up 15 months after inclusion.
  Immunological markers in blood identified in the on-going study ImmunoGraves Wp1 are analysed between participants who at follow up have 10.5 points or more at the Mental Fatigue Scale and participants who have less than 10.5 points at the Mental Fatigue Scale. Higher scores at the Mental Fatigue Scale means more brain fatigue.

SECONDARY OUTCOMES:
Levels of the previously identified immunological markers in serum at inclusion compared between participants who at follow up have high scores at the Mental Fatigue Scale and participants who at follow up have low scores at the Mental Fatigue Scale | Blood drawn at inclusion. Mental Fatigue Scale completed by participants at follow-up 15 months after inclusion.
  Immunological markers identified in the on-going study ImmunoGraves Wp1 are compared between participants who at follow up have 10.5 points or more at the Mental Fatigue Scale and participants who have less than 10.5 points at the Mental Fatigue Scale.Higher scores at the Mental Fatigue Scale means more brain fatigue.
Levels of the previously identified immunological markers in cerebrospinal fluid at inclusion compared between patients with high and low scores at the Mental Fatigue Score at follow-up | Cerebrospinal fluid drawn at inclusion. Mental Fatigue Scale completed by participants at follow-up 15 months after inclusion
  Immunological markers identified in the on-going study ImmunoGraves Wp1 are compared between participants who at follow up have 10.5 points or more at the Mental Fatigue Scale and participants who have less than 10.5 points at the Mental Fatigue Scale.Higher scores at the Mental Fatigue Scale means more brain fatigue.
Levels of the previously identified immunological markers in serum at follow up compared between patients with high and low scores at the Mental Fatigue Scale at follow-up and to healthy controls | Blood drawn and Mental Fatigue Scale completed by participants at follow-up 15 months after inclusion.
  Immunological markers identified in the on-going study ImmunoGraves Wp1 are compared between participants who at follow-up have 10.5 points or more at the Mental Fatigue Scale and participants who have less than 10.5 points at the Mental Fatigue Scale. Higher scores at the Mental Fatigue Scale means more brain fatigue.
Levels of the previously identified immunological markers in cerebrospinal fluid at follow up compared between patients with high and low scores at the Mental Fatigue Scale at follow-up | Cerebrospinal fluid drawn and Mental Fatigue Scale completed by participants at follow-up 15 months after inclusion.
  Immunological markers identified in the on-going study ImmunoGraves Wp1 are compared between participants who at follow-up have 10.5 points or more at the Mental Fatigue Scale and participants who have less than 10.5 points at the Mental Fatigue Scale. Higher scores at the Mental Fatigue Scale means more brain fatigue.
Levels of thyroid hormones at inclusion compared in patients with high and low scores at the Mental Fatigue Scale at follow-up | Blood drawn at inclusion. Mental Fatigue Scale completed by participants at follow-up 15 months after inclusion.
  Levels of thyroid hormones, analysed with the standard method of the laboratory at Sahlgrenska University Hospital, compared between participants who at follow-up have 10.5 points or more at the Mental Fatigue Scale and participants who have less than 10.5 points at the Mental Fatigue Scale. Higher scores at the Mental Fatigue Scale means more brain fatigue.
Levels of thyroid hormones at inclusion compared in patients with high and low scores at the Mental Fatigue Scale at inclusion | Blood drawn at inclusion. Mental Fatigue Scale completed by participants at inclusion.
  Levels of thyroid hormones, analysed with the standard method of the laboratory at Sahlgrenska University Hospital, compared between participants who at inclusion have 10.5 points or more at the Mental Fatigue Scale and participants who have less than 10.5 points at the Mental Fatigue Scale. Higher scores at the Mental Fatigue Scale means more brain fatigue.
Levels of thyroid antibodies at inclusion compared in patients with high and low scores at the Mental Fatigue Scale at follow-up | Blood drawn at inclusion. Mental Fatigue Scale completed by participants at follow-up 15 months after inclusion.
  Levels of thyroid autoantibodies, analysed with the standard method of the laboratory at Sahlgrenska University Hospital, compared between participants who at follow-up have 10.5 points or more at the Mental Fatigue Scale and participants who have less than 10.5 points at the Mental Fatigue Scale.Higher scores at the Mental Fatigue Scale means more brain fatigue.
Levels of thyroid antibodies at inclusion compared in patients with high and low scores at the Mental Fatigue Scale at inclusion | Blood drawn at inclusion. Mental Fatigue Scale completed by participants at inclusion.
  Levels of thyroid autoantibodies, analysed with the standard method of the laboratory at Sahlgrenska University Hospital, compared between participants who have 10.5 points or more at the Mental Fatigue Scale and participants who have less than 10.5 points at the Mental Fatigue Scale at inclusion. Higher scores at the Mental Fatigue Scale means more brain fatigue.
Levels of thyroid antibodies at follow-up compared in patients with high and low scores at the Mental Fatigue Scale at follow-up. | Blood drawn and Mental Fatigue Scale completed by participants at follow-up 15 months after inclusion.
  Levels of thyroid autoantibodies, analysed with the standard method of the laboratory at Sahlgrenska University Hospital, compared between participants who at follow-up have 10.5 points or more at the Mental Fatigue Scale and participants who have less than 10.5 points at the Mental Fatigue Scale.Higher scores at the Mental Fatigue Scale means more brain fatigue.
Levels of biomarkers indicating organic and structural nerve damage at inclusion in patients with high and low scores at the Mental Fatigue Scale at follow-up | Blood and, in a subgroup, cerebrospinal fluid drawn at inclusion. Mental Fatigue Scale completed by participants at follow-up 15 months after inclusion.
  Levels of biomarkers indicating organic and structural nerve damage, analysed with the standard method of the laboratory at Sahlgrenska University Hospital, compared between participants who at follow-up have 10.5 points or more at the Mental Fatigue Scale and participants who have less than 10.5 points at the Mental Fatigue Scale. Higher scores at the Mental Fatigue Scale means more brain fatigue.
Levels of biomarkers indicating organic and structural nerve damage at inclusion in patients with high and low scores at the Mental Fatigue Scale at inclusion | Blood and, in a subgroup, cerebrospinal fluid, drawn at inclusion. Mental Fatigue Scale completed by participants at inclusion.
  Levels of biomarkers indicating organic and structural nerve damage, analysed with the standard method of the laboratory at Sahlgrenska University Hospital, compared between participants who at inclusion have 10.5 points or more at the Mental Fatigue Scale and participants who have less than 10.5 points at the Mental Fatigue Scale. Higher scores at the Mental Fatigue Scale means more brain fatigue.
Levels of biomarkers indicating organic and structural nerve damage at follow-up in patients with high and low scores at the Mental Fatigue Scale at follow-up | Blood and, in a subgroup, cerebrospinal fluid, drawn at follow-up after 15 months. Mental Fatigue Scale completed by participants at follow-up 15 months after inclusion.
  Levels of biomarkers indicating organic and structural nerve damage, analysed with the standard method of the laboratory at Sahlgrenska University Hospital, compared between participants who at follow up have 10.5 points or more at the Mental Fatigue Scale and participants who have less than 10.5 points at the Mental Fatigue Scale.Higher scores at the Mental Fatigue Scale means more brain fatigue.
Prevalence of endocrine ophthalmopathy at inclusion compared between patients with high and low scores at the Mental Fatigue Scale at follow-up | Patients examined at inclusion, Mental Fatigue Scale completed by participants at follow-up 15 months after inclusion.
  Endocrine ophthalmopathy defined as Clinical Activity Score of 3/7 or more, compared between participants who at follow up have 10.5 points or more at the Mental Fatigue Scale and participants who have less than 10.5 points at the Mental Fatigue Scale. Higher scores at the Mental Fatigue Scale means more brain fatigue.
  Higher scores at the Clinical Activity Score means more serious endocrine ophthalmopathy.
Prevalence of endocrine ophthalmopathy at follow-up compared between patients with high and low scores at the Mental Fatigue Scale at follow-up | Patients examined and Mental Fatigue Scale completed by participants at follow-up 15 months after inclusion.
  Endocrine ophthalmopathy defined as Clinical Activity Score of 3/7 or more, compared between participants who at follow-up have 10.5 points or more at the Mental Fatigue Scale and participants who have less than 10.5 points at the Mental Fatigue Scale. Higher scores at the Mental Fatigue Scale means more brain fatigue. Higher scores at the Clinical Activity Score means more serious endocrine ophthalmopathy.
Scores at the Mental Fatigue Scale at inclusion compared between patients with Graves' with and without mental fatigue at follow-up and to healthy controls | Mental Fatigue Scale completed by participants at inclusion and follow-up at 15 months after inclusion, by controls at inclusion.
  Scores at the Mental Fatigue Scale at inclusion compared between participants who at follow-up have 10.5 points or more at the Mental Fatigue Scale and participants who have less than 10.5 points at the Mental Fatigue Scale. Higher scores at the Mental Fatigue Scale means more brain fatigue.
Self-evaluated quality of life in relation to ophthalmopathy compared between patients with Graves' with and without mental fatigue at follow-up, and to healthy controls. | Graves' Ophthalmopathy Quality of Life Questionnaire and Mental Fatigue Scale completed by participants at inclusion and follow-up at 15 months after inclusion, by controls at inclusion.
  Evaluated by the validated questionnaire the Graves' Ophthalmopathy Quality of Life Questionnaire (GO QoL). Scores are compared between participants who at follow-up have 10.5 points or more at the Mental Fatigue Scale and participants who have less than 10.5 points at the Mental Fatigue Scale. Higher scores at the Mental Fatigue Scale means more brain fatigue. Higher scores at the Graves' Ophthalmopathy Quality of Life Questionnaire means better quality of life.
Self-evaluated quality of life in relation to thyroid symptoms will be compared between patients with Graves' with and without mental fatigue at follow-up, and to healthy controls. | Thyroid-specific Patient-Reported Outcome short-form and Mental Fatigue Scale completed by participants at inclusion and follow-up 15 months after inclusion, by controls at inclusion.
  Evaluated by the validated questionnaire Thyroid-specific Patient-Reported Outcome short-form (ThyPro 39). Scores are compared between participants who at follow-up have 10.5 points or more at the Mental Fatigue Scale and participants who have less than 10.5 points at the Mental Fatigue Scale. Higher scores at the Mental Fatigue Scale means more brain fatigue.Higher scores at the Thyroid-specific Patient-Reported Outcome short-form means worse quality of life.
Self-evaluated quality of life and well-being will be compared between patients with Graves' with and without mental fatigue at follow-up and to healthy controls | Psychological General Well Being indexed Mental Fatigue Scale completed by participants at inclusion and follow-up 15 months after inclusion, by controls at inclusion.
  Evaluated by the validated questionnaire Psychological General Well Being index (PGWB). Scores are compared between participants who at follow-up have 10.5 points or more at the Mental Fatigue Scale and participants who have less than 10.5 points at the Mental Fatigue Scale. Higher scores at the Mental Fatigue Scale means more brain fatigue. Higher scores at the Psychological General Well Being means higher quality of life.
Self-evaluated symptoms of anxiety and depression compared between patients with Graves' with and without mental fatigue at follow-up and to healthy controls | Comprehensive Psychopathological Rating Scale and Mental Fatigue Scale completed by participants at inclusion and follow-up 15 months after inclusion, by controls at inclusion.
  Evaluated by the validated questionnaire the Comprehensive Psychopathological Rating Scale (CPRS). Scores are compared between participants who at follow-up have 10.5 points or more at the Mental Fatigue Scale and participants who have less than 10.5 points at the Mental Fatigue Scale. Higher scores at the Mental Fatigue Scale means more brain fatigue. Higher scores at the Comprehensive Psychopathological Rating Scale mean more symptoms of anxiety and depression.
Self-evaluated stress compared between patients with Graves' with and without mental fatigue at follow-up and to healthy controls | Perceived Stress Scale and Mental Fatigue Scale completed by participants at inclusion and follow up 15 months after inclusion, by controls at inclusion.
  Evaluated by the validated questionnaire Perceived Stress Scale (PSS-14). Scores are compared between participants who at follow-up have 10.5 points or more at the Mental Fatigue Scale and participants who have less than 10.5 points at the Mental Fatigue Scale. Higher scores at the Perceived Stress Scale mean more symptoms of stress.
Coping strategies will be compared between patients with Graves' with and without mental fatigue at follow-up, and to healthy controls | Brief cope and Mental Fatigue Scale completed by participants at inclusion and follow up 15 months after inclusion, by controls at inclusion.
  Evaluated by the validated questionnaire Brief cope. Coping strategies are compared between participants who at follow-up have 10.5 points or more at the Mental Fatigue Scale and participants who have less than 10.5 points at the Mental Fatigue Scale.
Optimistic self-beliefs to cope with difficulties in life will be compared between patients with Graves' with and without mental fatigue at follow-up and to healthy controls. | General self efficacy and Mental Fatigue Scale completed by participants at inclusion and follow-up 15 months after inclusion, by controls at inclusion.
  Evaluated by the validated questionnaire General Self-Efficacy. Scores are compared between participants who at follow-up have 10.5 points or more at the Mental Fatigue Scale and participants who have less than 10.5 points at the Mental Fatigue Scale. Higher scores at the General Self-Efficacy questionnaire means higher optimistic self-beliefs.
Personality traits will be compared between patients with Graves' with and without mental fatigue at follow-up, and to healthy controls | NEO Five-Factor Inventory-3 and Mental Fatigue Scale completed by participants at inclusion and follow-up 15 months after inclusion, by controls at inclusion.
  Evaluated by the validated questionnaire NEO Five-Factor Inventory-3 (NEO-FFI-3). Personality traits are compared between participants who at follow-up have 10.5 points or more at the Mental Fatigue Scale and participants who have less than 10.5 points at the Mental Fatigue Scale.
Observations of hippocampal neuronal activation during attention testing in hyperthyroidism and in healthy controls. | Magnetoencephalography will be performed in patients and in controls at inclusion.
  Magnetoencephalography will be performed in a subset of patients and in healthy controls. Combined with magneto resonance imaging (MRI), magnetoencephalography gives information on neuronal activation by measuring alfa- and theta-band oscillations during attention testing.
Observations of neuronal activation during attention testing in patients with Graves' disease at follow-up and in healthy controls. | Magnetoencephalography will be performed in patients at follow-up 15 months after inclusion, in controls at inclusion.
  Magnetoencephalography will be performed in a subset of patients and in healthy controls. Combined with magneto resonance imaging (MRI), magnetoencephalography gives information on neuronal activation by measuring alfa- and theta-band oscillations during attention testing.
Observations of neuronal activation during attention testing at follow-up compared between patients with and without mental fatigue and in healthy controls. | Magnetoencephalography will be performed in patients after 15 months, in controls at inclusion. Mental Fatigue Scale will be completed by patients at follow-up 15 months after inclusion, by controls at inclusion.
  Magnetoencephalography will be performed in a subset of patients and in healthy controls. Combined with magneto resonance imaging (MRI), magnetoencephalography gives information on neuronal activation by measuring alfa- and theta-band oscillations during attention testing. The alfa- and theta-band oscillations will be compared between participants who at follow-up have 10.5 points or more at the Mental Fatigue Scale and participants who have less than 10.5 points at the Mental Fatigue Scale.
Immunological markers from Primary Outcome will be compared in patients with changed hippocampal neuronal activation compared to controls, and in controls. | Magnetoencephalography will be performed in patients at inclusion and after 15 month, in controls at inclusion. Blood and cerebrospinal fluid will be drawn at inclusion.
  Magnetoencephalography will be performed in a subset of patients and in healthy controls. Combined with magneto resonance imaging (MRI), magnetoencephalography gives information on neuronal activation by measuring alfa- and theta-band oscillations during attention testing. Immunological markers identified in the on-going study ImmunoGraves wp1 and in Primary Outcome.
Immunological markers from Primary Outcome will be compared in patients without changed hippocampal neuronal activation compared to controls, and in controls. | Magnetoencephalography will be performed in patients at inclusion and after 15 months, in controls at inclusion. Blood and cerebrospinal fluid will be drawn at inclusion.
  Magnetoencephalography will be performed in a subset of patients and in healthy controls. Combined with magneto resonance imaging (MRI), magnetoencephalography gives information on neuronal activation by measuring alfa- and theta-band oscillations during attention testing. Immunological markers identified in the on-going study ImmunoGraves wp1 and in Primary Outcome.
Biomarkers indicating organic and structural nerve damage will be compared in patients without changed hippocampal neuronal activation compared to controls, and in controls. | Magnetoencephalography will be performed in patients at inclusion and at follow-up 15 months after inclusion, in controls at inclusion. Blood and cerebrospinal fluid will be drawn at inclusion.
  Magnetoencephalography will be performed in a subset of patients and in healthy controls. Combined with magneto resonance imaging (MRI), magnetoencephalography gives information on neuronal activation by measuring alfa- and theta-band oscillations during attention testing. Biomarkers indicating organic and structural nerve damage analysed with the standard method of the laboratory at Sahlgrenska University Hospital.
Thyroid autoantibodies will be compared in patients with changed hippocampal neuronal activation compared to controls, and in controls. | Magnetoencephalography will be performed in patients at inclusion and after 15 months, in controls at inclusion. Blood and cerebrospinal fluid will be drawn at inclusion.
  Magnetoencephalography will be performed in a subset of patients and in healthy controls. Combined with magneto resonance imaging (MRI), magnetoencephalography gives information on neuronal activation by measuring alfa- and theta-band oscillations during attention testing. Thyroid autoantibodies analysed with the standard method of the laboratory at Sahlgrenska University Hospital.
Thyroid autoantibodies will be compared in patients without changed hippocampal neuronal activation compared to controls, and in controls. | Magnetoencephalography will be performed in patients at inclusion and after 15 months, in controls at inclusion. Blood and cerebrospinal fluid will be drawn at inclusion.
  Magnetoencephalography will be performed in a subset of patients and in healthy controls. Combined with magneto resonance imaging (MRI), magnetoencephalography gives information on neuronal activation by measuring alfa- and theta-band oscillations during attention testing. Thyroid autoantibodies analysed with the standard method of the laboratory at Sahlgrenska University Hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Filipsson, ass prof, Principal Investigator — Institute of Medicine, Sahlgrenska Academy, University of Gothenburg, Department of Endocrinology, Sahlgrenska University Hospital, Wallenberg Center for Molecular and Translational Medicine, all in Gothenburg, Sweden
Locations (1):
- Endokrina Forskningsenheten, Sahlgrenska University Hospital, Gothenburg, Sweden